CLINICAL TRIAL: NCT02091778
Title: Open, Non-comparative, Multi-centre Post Marketing Clinical Follow-up Investigation to Evaluate Performance and Safety on Diabetic Foot Ulcer, DFU When Using Fast Gelling Dressing as Intended.
Acronym: CHEXU 01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEXU 01
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fast Gelling Dressing (Experimental)
  Interventions: Device: Fast gelling dressing

INTERVENTIONS:
Device: Fast gelling dressing

SUMMARY:
The primary objective of this post market clinical follow-up (PMCF) investigation is to evaluate performance and safety of fast gelling dressing when used as intended in Diabetic Foot Ulcer (DFU).

The primary endpoint will be Changes from baseline in the condition of the peri-wound skin measured by the following variables; maceration, redness/irritation, rash/eczema, blistering, dermatitis, skin stripping, trauma to wound edges and product degradation on the skin

ELIGIBILITY:
Inclusion Criteria:

1. Both gender ≥18 years old.
2. Subjects with type 1 or 2 diabetes mellitus.
3. Texas Grade A1 or 2, C1 or 2
4. Exuding diabetic foot ulcer
5. Ulcer localisation; below the ankle
6. Signed Informed Consent.

Exclusion Criteria:

1. Known allergy/hypersensitivity to the dressing.
2. HbA1c ≥ 10% (86 mmol/mol) (most recent value within 3 months)
3. Wound infection requiring systemic treatment
4. Subjects who will have problems following the protocol.
5. Subjects included in other ongoing clinical investigation at present or during the past 30 days.
6. Toe pressure less than 70 mmHg
7. Clinical suspicion of osteomyelitis (based on probe to bone/radiological changes)
8. Dry wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Salford Royal Hospital (NHS) Foundation Trust, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- Fast Gelling Dressing: Fast gelling dressing
Period: Overall Study
Arm/Group | Fast Gelling Dressing
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fast Gelling Dressing
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Peri-wound Skin
Description: Measured by the following variables; maceration, redness/irritation, rash/eczema, blistering, dermatitis, skin stripping, trauma to wound edges and product degradation on the skin
Time Frame: 12 weeks
Population: number of patients with healthy/intact peri-wound skin that increased from baseline to final visit. (From 6 to 14)
Measure: Number; unit: participants
Arm/Group | Fast Gelling Dressing
Number analyzed (Participants) | 21
participants | 8

ADVERSE EVENTS:
Arm/Group | Fast Gelling Dressing
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast Gelling Dressing (N=21)
abdominal pain & pain in abdomen. (Endocrine disorders) | 2 (2) — abdominal pain & pain in abdomen.
high temperature and un-well, (Infections and infestations) | 1 (1) — high temperature and un-well,
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast Gelling Dressing (N=21)
Infection to ulcer site, (Infections and infestations) | 1 (1) — Infection to ulcer site,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No